CLINICAL TRIAL: NCT01746914
Title: Morphofunctional Lung Analysis by Positron Emission Tomography and Computed Tomography After Lung Transplantation
Brief Title: Morphofunctional Lung Analysis by PET and CT After Lung Transplantation
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Other Study IDs: 201212
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Disorder Related to Lung Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung transplantated patients: Patients undergone lung transplantation

SUMMARY:
72 hours after lung transplantation, patients undergo a positron emission tomography (PET) scan and a computed tomography (CT) scan in order to analyse lung function and morphology.

Aim of the study is to analyse complications onset (in particular primary graft dysfunction), and evaluate 90 days mortality after lung transplantation.

DETAILED DESCRIPTION:
Pulmonary transplantation is considered as a lifesaving procedure in end-stage pulmonary disease. However morbidity and mortality after lung transplantation are still significant.

Primary graft dysfunction (PGD) is the main cause of early death. PGD is similar to acute lung injury (ALI)/ acute respiratory distress syndrome (ARDS): oxygenation is compromised, pulmonary compliance is decreased, chest Rx shows several infiltrates, and alveolar damage is present.

25% of patients develops PGD within 72 hours from transplantation and 30 days mortality is eight times higher in patients who develop PGD.

72 hours after lung transplantation, patients, whose clinical condition allow to bring them to nuclear medicine department, will undergo pulmonary computed tomography (CT) to study lung morphology and measure lung recruitability and positron emission tomography (PET) to study lung functionality and estimate lung inflammation.

Aim of this study is to investigate the onset of PGD and other complications and to determine 72 hours and 90 days mortality after lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* lung transplantation
* ≥ 18 years

Exclusion Criteria:

* < 18 years
* patient' s clinical conditions not allowing patient transport from ICU to Nuclear Medicine Unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung Transplantated patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of patients alive | up to 90 days from transplantation

SECONDARY OUTCOMES:
incidence of complications other than primary graft dysfunction | 72 hours and 90 days
incidence of primary graft dysfunction | 72 hours and 90 days after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Policlinico Hospital; Franco Valenza, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided